CLINICAL TRIAL: NCT02620085
Title: Bio-psycho-social Correlates of Psychological Distress in Patients With Graves' Disease in Euthyroid Status
Brief Title: Thyroid Disease and Personality Study
Acronym: TPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201107013RC
Record Dates: First submitted 2015-11-04; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Graves' Disease
Keywords: Graves' disease; Hyperthyroidism; Personality traits
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Graves' disease: Patient had been diagnosed of Graves' disease and now under euthyroid status
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — blood sampling

SUMMARY:
Observe the relationship between thyroid function and personality traits

DETAILED DESCRIPTION:
Thyrotoxicosis was the biochemical and physiological manifestations of excess thyroid hormone. The clinical manifestation was palpitation, heat intolerance, hand tremor, and weight loss. The clinical manifestation also included nervous system, including anxiety, tension, irritability, hyperactivity, fatigue, and insomnia.

Where tensions features include restless, short attention span, and the impulse to want to move around. Some patients will progress to a non-specific psychiatric disorders. According to the study, about 10% of patients will occur very frank psychosis, 3, 31% to 69% of patients with depressive symptoms, 61% to 62% of patients with symptoms of anxiety.

Some studies using reliable evaluation tool to evaluate behavioral changes in patients with thyrotoxicosis, such as Clyde emotional scale, multi-faceted personality assessment table (Multiphasic Personality Inventory (MMPI)), or observation of a response time to visual or audio stimulation. After treatment of thyrotoxicosis, most of these indicators have improved, but some indicators were still abnormal after treatment of thyrotoxicosis, such as MMPI and voice response time.

The physiological causes of the changes of these nervous system is not clear. The symptoms was improved after the use of sympathetic inhibitors, so presumably this may correlated with autonomic nervous system disorders.

Thyroid hormone receptors are widely distributed in the brain may also be one of the cause. But there still some other reasons for the changes of neurological symptoms because neurological symptoms may not be back to normal even after thyroid function returned to normal. Autoimmune dysfunction affect brain function may be the most possible reason. Graves' disease is the most common cause of thyrotoxicosis and it is related to autoimmune thyroid antibodies.

Clinically, some patients of Graves' disease may combined with other autoimmune disease, such as Sicca syndrome. The patient may still have nervous personality traits despite normalized thyroid function. Some patients even need long-term use of anti-anxiety medication.

In this study, investigators hope to analyze the personality traits of patients with hyperthyroidism,especially patients of Graves' disease, in Taiwan and to observe the changes during treatment. Investigators also hope to observe the statistical change of other non-thyroid-specific autoimmune index in this thyrotoxicosis patient. After obtaining these results, investigators will evaluate whether to continue to study the hypothesis of affection of brain of thyrotoxic patients by the abnormal autoimmune system.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 85 years
* euthyroid Graves' disease

Exclusion Criteria:

* Patients who were not capable to complete the questionnaire due to severe cognitive dysfunction or under education were excluded from this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were aged between 20 and 85 years and fulfilled the criteria for euthyroid GD. GD is defined by a history of hyperthyroidism, thyroid eye disease or pretibial myxedema with abnormal high thyroglobulin binding immunoglobulin (TBII) level and autoimmune characteristics on thyroid echography. Euthyroidism is defined by normal free thyroxine (fT4) and thyrotropin (TSH) level.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Psychological distress in scores measured using the Brief Symptom Rating Scale | Within one year after inclusion
  Psychological distress is measured by using the Brief Symptom Rating Scale (BSRS). The BSRS is a self-report questionnaire with 30 items rated from 0 to 4 scores on the basis of the degree of distress. BSRS covers nine dimensions of psychopathology: somatization, obsessive-compulsive disorder, interpersonal sensitivity, depression, anxiety, hostility, phobic-anxiety, paranoid ideation, and additional symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- Shyang-Rong Shih, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Kathol RG, Delahunt JW. The relationship of anxiety and depression to symptoms of hyperthyroidism using operational criteria. Gen Hosp Psychiatry. 1986 Jan;8(1):23-8. doi: 10.1016/0163-8343(86)90060-5. PMID 3943712
- [Background] Trzepacz PT, McCue M, Klein I, Levey GS, Greenhouse J. A psychiatric and neuropsychological study of patients with untreated Graves' disease. Gen Hosp Psychiatry. 1988 Jan;10(1):49-55. doi: 10.1016/0163-8343(88)90084-9. PMID 3345907
- [Background] BURSTEN B. Psychoses associated with thyrotoxicosis. Arch Gen Psychiatry. 1961 Mar;4:267-73. doi: 10.1001/archpsyc.1961.01710090053007. No abstract available. PMID 13689243
- [Background] Lee MB, Lee YJ, Yen LL, Lin MH, Lue BH. Reliability and validity of using a Brief Psychiatric Symptom Rating Scale in clinical practice. J Formos Med Assoc. 1990 Dec;89(12):1081-7. PMID 1982678
- [Background] Lee YC, Wang HP, Chiu HM, Liao SC, Huang SP, Lai YP, Wu MS, Chen MF, Lin JT. Comparative analysis between psychological and endoscopic profiles in patients with gastroesophageal reflux disease: a prospective study based on screening endoscopy. J Gastroenterol Hepatol. 2006 May;21(5):798-804. doi: 10.1111/j.1440-1746.2005.04034.x. PMID 16704526
- [Background] Liao SC, Lee MB, Lee YJ, Huang TS. Hyperleptinemia in subjects with persistent partial posttraumatic stress disorder after a major earthquake. Psychosom Med. 2004 Jan-Feb;66(1):23-8. doi: 10.1097/01.psy.0000106880.22867.0e. PMID 14747634
- [Background] Chen CA, Liao SC, Wang JK, Chang CI, Chiu IS, Chen YS, Lu CW, Lin MT, Chiu HH, Chiu SN, Hua YC, Lue HC, Wu MH. Quality of life in adults with congenital heart disease: biopsychosocial determinants and sex-related differences. Heart. 2011 Jan;97(1):38-43. doi: 10.1136/hrt.2010.200709. Epub 2010 Oct 26. PMID 20978017
- [Background] Hsu YC, Liou JM, Liao SC, Yang TH, Wu HT, Hsu WL, Lin HJ, Wang HP, Wu MS. Psychopathology and personality trait in subgroups of functional dyspepsia based on Rome III criteria. Am J Gastroenterol. 2009 Oct;104(10):2534-42. doi: 10.1038/ajg.2009.328. Epub 2009 Jun 16. PMID 19532128
- [Background] Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. Psychopharmacol Bull. 1973 Jan;9(1):13-28. No abstract available. PMID 4682398
- [Background] Liao SC, Lee MB, Lee YJ, Weng T, Shih FY, Ma MH. Association of psychological distress with psychological factors in rescue workers within two months after a major earthquake. J Formos Med Assoc. 2002 Mar;101(3):169-76. PMID 12051011
- [Background] Lee MB, Rin H, Lin HN, Lee YJ Personality as an effective predictor of outcome for neurotic disorders. Chinese Psychiatry 1990; 4:111-121.
- [Background] BARTHOLOMEW AA, MARLEY E. The temporal reliability of the Maudsley personality inventory. J Ment Sci. 1959 Jan;105(438):238-40. doi: 10.1192/bjp.105.438.238. No abstract available. PMID 13641975
- [Background] EYSENCK HJ. Personality. Annu Rev Psychol. 1952;3:151-74. doi: 10.1146/annurev.ps.03.020152.001055. No abstract available. PMID 12977189
- [Background] Smilkstein G, Ashworth C, Montano D. Validity and reliability of the family APGAR as a test of family function. J Fam Pract. 1982 Aug;15(2):303-11. PMID 7097168
- [Background] Schreckenberger MF, Egle UT, Drecker S, Buchholz HG, Weber MM, Bartenstein P, Kahaly GJ. Positron emission tomography reveals correlations between brain metabolism and mood changes in hyperthyroidism. J Clin Endocrinol Metab. 2006 Dec;91(12):4786-91. doi: 10.1210/jc.2006-0573. Epub 2006 Sep 12. PMID 16968792
- [Background] Jaracz J, Kucharska A, Rajewska-Rager A, Lacka K. Cognitive functions and mood during chronic thyrotropin-suppressive therapy with L-thyroxine in patients with differentiated thyroid carcinoma. J Endocrinol Invest. 2012 Sep;35(8):760-5. doi: 10.3275/8013. Epub 2011 Oct 6. PMID 21986400
- [Background] Boelaert K, Newby PR, Simmonds MJ, Holder RL, Carr-Smith JD, Heward JM, Manji N, Allahabadia A, Armitage M, Chatterjee KV, Lazarus JH, Pearce SH, Vaidya B, Gough SC, Franklyn JA. Prevalence and relative risk of other autoimmune diseases in subjects with autoimmune thyroid disease. Am J Med. 2010 Feb;123(2):183.e1-9. doi: 10.1016/j.amjmed.2009.06.030. PMID 20103030
- [Background] Kirshner HS. Hashimoto's encephalopathy: a brief review. Curr Neurol Neurosci Rep. 2014 Sep;14(9):476. doi: 10.1007/s11910-014-0476-2. PMID 25027262
- [Derived] Lin CH, Chang CK, Shih CW, Li HY, Chen KY, Yang WS, Tsai KS, Wang CY, Shih SR. Serum fibroblast growth factor 23 and mineral metabolism in patients with euthyroid Graves' diseases: a case-control study. Osteoporos Int. 2019 Nov;30(11):2289-2297. doi: 10.1007/s00198-019-05116-1. Epub 2019 Aug 5. PMID 31384956